CLINICAL TRIAL: NCT06388382
Title: Investigation of the Audible Alert Tone in ICD Patients with Subcutaneous Cardioverter Defibrillators
Brief Title: Investigation of the Audible ICD Alert Tone
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Other Study IDs: UKKx2024
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Implantable Defibrillator User

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Alert tone demonstration — Patients are demonstrated the alert tone of their ICD

SUMMARY:
Ability of ICD patients to hear the audible ICD alert is being assessed.

ELIGIBILITY:
Inclusion Criteria:

* patient equipped with a subcutaneous ICD
* willing to participate

Exclusion Criteria:

* S-ICD implantation within the past 3 weeks
* patient is deaf

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: S-ICD all comers
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Alert tone audible | 1 minute after demonstration
  Patients state if they hear or don't hear the alert tone

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided